CLINICAL TRIAL: NCT06967974
Title: Evaluation of Tai Chi for Chronic Insomnia Disorder Combined With Hyperarousal/Anxiety
Brief Title: Effects of Tai Chi on Chronic Insomnia Disorder Combined With Hyperarousal/Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tai Chi for CI
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Chronic Insomnia
Keywords: Chronic Insomnia; Tai Chi; hyperawareness; anxiety
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai Chi + Sleep Hygiene Education (Experimental)
  Interventions: Other: Tai Chi + Sleep Hygiene Education
- Sleep Hygiene Education (Active Comparator)
  Interventions: Other: Sleep Hygiene Education

INTERVENTIONS:
Other: Tai Chi + Sleep Hygiene Education — Conduct simplified training on the 24 style Tai Chi; Sleep hygiene education includes adjusting sleep time, maintaining regular lifestyle habits, optimizing bedroom environment, reducing nighttime stimulation, avoiding thinking when going to bed, adjusting alarm clock positions, and reducing daytime napping.
  Arms: Tai Chi + Sleep Hygiene Education
Other: Sleep Hygiene Education — Participants will receive Sleep Hygiene Education, consisting of guidance on establishing healthy sleep habits, optimizing sleep environment, adjusting sleep schedules, reducing stimulants (e.g., caffeine, alcohol), and minimizing sleep-disruptive behaviors.
  Arms: Sleep Hygiene Education

SUMMARY:
This study focuses on individuals with chronic insomnia combined with excessive arousal/anxiety, with the main objective of investigating the effectiveness of Tai Chi in treating CI with excessive arousal/anxiety.

DETAILED DESCRIPTION:
Patients with chronic insomnia often experience both daytime fatigue and difficulty falling asleep at night, as well as shallow sleep and easy awakening, which is a manifestation of 24-hour excessive wakefulness. Additionally, insomnia is often associated with anxiety and tension. Therefore, for patients with chronic insomnia accompanied by anxiety, relieving anxiety is often an important means of treating insomnia. In recent years, an increasing number of studies have shown that Tai Chi has potential therapeutic value in treating mental disorders such as insomnia and anxiety. Tai Chi is a coordinated and unified physical and mental exercise that regulates the body's functional state through rhythmic and regular physical activities, and is combined with psychological "relaxation" activities. Therefore, the investigators propose the hypothesis that Tai Chi training may improve chronic insomnia with excessive arousal/anxiety through intermediate pathways such as neuroendocrine, immune function, neurochemistry, etc. This study aims to explore the effects of Tai Chi on chronic insomnia combined with excessive arousal/anxiety, broaden new ideas for non pharmacological treatment of sleep problems, and provide data reference for the development of more precise sleep aid exercise plans in the future.

ELIGIBILITY:
Inclusion Criteria:

1. meet DSM-5 diagnostic criteria for insomnia disorder;
2. Pittsburgh Sleep Quality Index (PSQI) total score >5;
3. age ≥18 years old with junior high school education or above;
4. voluntarily participate in this study by signing an informed consent form; and 5) HAMA ≥14 was required for those who had chronic insomnia disorder with anxiety symptoms.

Exclusion Criteria:

1. people with comorbid serious physical or severe mental illnesses, suicide risk;
2. clinically diagnosed or suspected sleep breathing disorder, restless legs syndrome and sleep-wake rhythm disorder, shift workers;
3. pregnant and breastfeeding women; and
4. people who are currently undergoing any psychological treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Difference in change from baseline in Pittsburgh sleep quality index (PSQI) scores at the end of treatment between the two groups. | Baseline to week 6

SECONDARY OUTCOMES:
Differences in the values of change from baseline in Hamilton Anxiety Scale (HAMA) scores at the end of treatment, and at 3 months, 6 months, and 12 months of follow-up between the two groups. | Baseline to week 6, month 3, month 6, and month 12
  The scale consists of 14 items, and each item is rated on a 5-point scale from 0-4, with a total score of ≥29 for probable severe anxiety, a total score of ≥21 for definite significant anxiety, a total score of ≥14 for definite anxiety, a total score of ≥7 for probable anxiety, and <7 for no symptoms of anxiety.
Differences in change from baseline in Beck Anxiety Inventory (BAI) scores at the end of treatment, and at 3 months, 6 months and 12 months of follow-up between the two groups. | Baseline to week 6, month 3, month 6, and month 12
  The scale contains 21 items and uses a 4-point scale method, with a total score of 15-25 as mild anxiety, 26-35 as moderate anxiety, and 36 or more as severe anxiety.
Differences in the change from baseline in the insomnia severity index (ISI) scores at the end of treatment and at 3, 6 and 12 months of follow-up between the two groups. | Baseline to week 6, month 3, month 6, and month 12
  The scale is divided into 7 sections with a total score of 0-28, with higher scores indicating more severe insomnia. The degree of insomnia is classified according to the scores: 0-7 indicates no insomnia, 8-14 is mild insomnia, 15-21 is moderate insomnia, and 22-28 is severe insomnia.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No